CLINICAL TRIAL: NCT05070234
Title: Genetic Diagnosis and the Response to Recombinant Human Growth Hormone Treatment in Small for Gestational Age Children With Short Stature
Brief Title: Genetic Diagnosis and Human Growth Hormone Treatment in Small for Gestational Age Children With Short Stature
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Chunxiu Gong (Other)
Collaborators: Shanghai Children's Hospital (Other); Second Affiliated Hospital of Guangzhou Medical University (Other); Shenzhen Children's Hospital (Other Government); Tongji Hospital (Other); The Children's Hospital of Zhejiang University School of Medicine (Other); Chengdu Women's and Children's Central Hospital (Other); West China Second University Hospital (Other); The First Affiliated Hospital with Nanjing Medical University (Other); Changchun GeneScience Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor-Investigator, Chunxiu Gong, Department of Endocrinology, Genetics and Metabolism, Beijing Children's Hospital
Organization: Beijing Children's Hospital (Other)
Other Study IDs: GenSci-GH-21016
Record Dates: First submitted 2021-09-27; First posted 2021-10-07 (Actual); Last update posted 2021-10-07 (Actual); Status verified 2021-09

CONDITIONS: Small for Gestational Age Infant; Silver-Russell Syndrome; Genetic Diseases, Inborn
MeSH Terms: conditions — Silver-Russell Syndrome; Genetic Diseases, Inborn | interventions — Genetic Testing

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — whole blood
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- short stature children born small for gestational age: This group was defined as a group of children whose birth weight and/or birth length equal or less than -2 SD for sex and gestational age, and who had failed to catch up in growth, remaining short after 2 years old.
  Interventions: Genetic: Blood collection for genetic analysis

INTERVENTIONS:
Genetic: Blood collection for genetic analysis — Genetic tests in this study are sequential testing, including MS-MLPA, whole exome sequencing, whole genome sequencing, as well as RNA-seq.

SUMMARY:
This study is a multi-center, retrospective and non-interventional research. In this study, a total of 150 short children who were small for gestational age and had been treated with recombinant human growth hormone (rhGH) are selected for genetic testing. The aims of this study are to analyze the genetic etiology of SGA children with short stature, and to compare the efficacy and safety of rhGH treatment in subjects with different etiologies.

ELIGIBILITY:
Inclusion Criteria:

1. Single birth, clinical diagnosis of SGA;
2. rhGH treatment beginned before puberty (Tanner stage I), regardless of gender;
3. Before starting rhGH treatment, height was lower than -2 SDS compared with normal children of the same age and sex;
4. All the subjects and their guardians signed the informed consent and the informed consent for genetic testing.

Exclusion Criteria:

1. No efficacy and safety data were recorded after treatment with rhGH;
2. A history of blood transfusion within 3 months before the collection of the genetic blood samples, or a history of bone marrow transplantation between rhGH treatment and the enrollment in this study;
3. Other conditions that the investigator considered unsuitable for inclusion in this study.

Ages: 2 Years to 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Children's hospical
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2021-10-11 (Estimated); Primary Completion 2022-08-30 (Estimated); Study Completion 2022-08-30 (Estimated)

PRIMARY OUTCOMES:
Genetic testing | At baseline
  To detect the disease-causing genes of SGA children with short stature

CONTACTS AND LOCATIONS:
Overall Officials: Chunxiu Gong, doctor, Principal Investigator — Beijing Children's Hospital

IPD SHARING:
Plan to Share IPD: No